CLINICAL TRIAL: NCT00013169
Title: Patient-Centered Alternative to Psychiatric Hospitalization for Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCC 98-051
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Veterans; Acute Hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Strong Patient Focus

INTERVENTIONS:
Behavioral: Strong Patient Focus

SUMMARY:
A variety of models of psychiatric hospital alternative care have been developed over the past several decades. San Diego�s Short-Term Acute Residential Treatment (START) model is one of the best established of these alternatives, comprising a network of 6 facilities with a total of 77 beds. Although veterans have been among those served at START programs for many years, no previous study of START or any other model has focused specifically on veterans.

DETAILED DESCRIPTION:
Background:

A variety of models of psychiatric hospital alternative care have been developed over the past several decades. San Diego�s Short-Term Acute Residential Treatment (START) model is one of the best established of these alternatives, comprising a network of 6 facilities with a total of 77 beds. Although veterans have been among those served at START programs for many years, no previous study of START or any other model has focused specifically on veterans.

Objectives:

The study tested the hypotheses that veterans treated in a START program would demonstrate greater improvement in symptoms and quality of life, as well as greater satisfaction with treatment and lower costs of care than veterans treated at the VA inpatient unit.

Methods:

This study includes elements of both efficacy and effectiveness studies. VA psychiatric unit treatment and START are compared in a randomized trial, with follow up of subjects at 2, 6, and 12 months as they experience real-world treatment-as-usual. Symptoms, functioning, quality of life, and satisfaction with services are assessed on multiple standardized measures, as well as by qualitative assessments.

Status:

Final report is under preparation.

ELIGIBILITY:
Inclusion Criteria:

Have to a veteran and in need of acute hospitalization, but able to take care of themselves. (Max Age is 59)

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Lohr, MD BA, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

REFERENCES:
- [Result] Ta S, Goldzweig C, Juzba M, Lee M, Wenger N, Yano EM, Asch S. Addressing physician concerns about performance profiling: experience with a local Veterans Affairs quality evaluation program. Am J Med Qual. 2009 Mar-Apr;24(2):123-31. doi: 10.1177/1062860608330828. Epub 2009 Feb 19. PMID 19228893